CLINICAL TRIAL: NCT00665184
Title: High Force Resistance Training and Dopamine Replacement Effects on Hypokinesia in Parkinson Disease
Brief Title: Strength Training and Medication Effects in Parkinson Disease Effects on Hypokinesia in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lee Dibble, Associate Professor, University of Utah
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 11900; 1R15HD056478-01 (NIH)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Parkinson Disease
Keywords: Hypokinesia; Gait; Quality of life; Dopamine replacement; Resistance training
MeSH Terms: conditions — Parkinson Disease; Hypokinesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High force LE resistance training (Experimental): High force lower extremity resistance training + Standard exercise care. The high force lower extremity resistance training group will participate in a 3 day per week progressive eccentric ergometry program that will be gradually increased over 3 weeks from 5-20 minutes per day and remain at that duration for the next 9 weeks. In addition, they will engage in exercises including moderate intensity aerobic training, concentric upper extremity resistance training and stretching (axial mobility exercises).
  Interventions: Behavioral: Resistance Exercise via Negative Eccentric Work
- Standard Care Control Group (Active Comparator): Standard care exercise group: The standard care control group is an "active control group", i.e., individuals who will engage in our standard of care (an evidence based exercise program). These exercises include moderate intensity aerobic training (15 minutes), concentric upper extremity resistance training (5-10 minutes), balance training (5 minutes), and stretching (axial mobility exercises-5-10 minutes).
  Interventions: Behavioral: Standard care exercise training

INTERVENTIONS:
Behavioral: Resistance Exercise via Negative Eccentric Work — High intensity resistance training delivered 2-3 times per week for 12 weeks
  Arms: High force LE resistance training
Behavioral: Standard care exercise training — Evidence based exercise training (resistance training, aerobic training, flexibility training) 2-3 times per week for 12 weeks.
  Arms: Standard Care Control Group

SUMMARY:
Parkinson disease is a degenerative neurologic condition characterized by slowness of movement, tremor, and loss of balance control. It results in significant degrees of disability for affected individuals. Exercise and medication management are two treatments frequently used to treat Parkinson disease, and although some individuals benefit from these treatments, by what effect exercise works is presently not known. We will examine muscle structure and movement control responses to strengthening exercises and compare them to the therapeutic response observed as a result of medication intake. This process will allow us to better understand the mechanisms underlying the therapeutic effects of strengthening exercise for persons with Parkinson disease.

DETAILED DESCRIPTION:
Idiopathic Parkinson disease (IPD) is the model movement disorder to explore the motor function of the basal ganglia. (Morris ME, 2005) Alterations in the output of the basal ganglia lead to reductions in muscle force output and movement amplitude while inactivity and impaired mobility contribute to the loss of muscle size and strength.

Collectively these factors lead to reductions in the size and speed (hypokinesia) of functional movements such as gait. Hypokinesia during gait initiation and gait are biomechanical events that can precipitates movement deficits such as bradykinesia and falls. Previous studies have suggested that resistance training is beneficial in the management of persons with PD. Although anatomic, behavioral, and mobility related improvements have been demonstrated with resistance training intervention, it is unclear if the observed changes are derived solely from peripheral musculoskeletal changes or from central nervous system mediated alterations in force output and movement amplitude. The responsiveness of muscle force, movement amplitude, and hypokinesia to the CNS mediated effects of dopamine replacement provide a model system to which the effects of resistance training can be compared. In order to examine this question, we plan to conduct a controlled trial to rigorously examine the effects of high force resistance training on muscle structure, muscle force output, and hypokinesia in persons with moderate IPD and in the process, characterize the potentially differential effects of resistance training effects and dopamine replacement. This study assembles a team of investigators with experience in high force resistance training, measurement of the biomechanical and clinical balance function in persons with PD, and the statistical analysis expertise. Persons with IPD will be recruited, examined, and if they meet the inclusion criteria will be randomly assigned to one of two groups (experimental or standard care control). A battery of tests including muscle structure, muscle force production, and measures of hypokinesia and will be assessed on and off dopamine replacement medication both prior to and after a 12 week resistance training intervention. The first specific aim of the study is to determine if high force resistance training results in improvements in muscle structure, muscle force output, and hypokinesia in persons with moderate IPD. The second specific aim is to characterize and compare any differential effects of high force resistance training and dopamine replacement on muscle force output and hypokinesia in persons with moderate IPD. We hypothesize that dopamine replacement and resistance training will interact to improve muscle force output and reduce hypokinesia. In addition, we hypothesize that examination of kinematic patterns during gait initiation will reveal differential effects on lower extremity hypokinesia. The results of this study will help to better understand the differential contributions of resistance training and dopamine replacement on hypokinesia in persons with PD.

ELIGIBILITY:
Inclusion Criteria:

male or a female at least 40 years of age or older neurologist diagnosed idiopathic PD (using UK Brain Bank Criteria) ambulatory and medically cleared by their physician to participate in an exercise regimen clinical signs of hypokinesia (reduced movement amplitude during ADL tasks) or postural instability have a Folstein Mini-Mental State Examination score > 23 currently taking dopamine replacement medication

Exclusion Criteria:

previous surgical management of PD (pallidotomy, DBS) motor fluctuations and or dyskinesias uncontrolled by medications. central nervous system disorder (e.g., other than Parkinson's disease) myopathic disease (e.g., focal myopathy) that affects skeletal muscle structure/function rheumatological disease that has an effect on muscle and/or mobility unstable cardiovascular disease that limits exercise abilities impaired knee flexion, <90 degrees, extreme claustrophobia (secondary to the inability to perform the MRI scans) regular (2-3x/week) aerobic or resistance exercise performed over the past 6 months

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Hypokinesia as measured by movement kinematics and kinetics | Pre intervention and post intervention

SECONDARY OUTCOMES:
Functional mobility as measured by gait / balance | Pre intervention and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dibble, PhD, PT, Principal Investigator — University of Utah Department of Physical Therapy
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Dibble LE, Hale T, Marcus RL, Gerber JP, Lastayo PC. The safety and feasibility of high-force eccentric resistance exercise in persons with Parkinson's disease. Arch Phys Med Rehabil. 2006 Sep;87(9):1280-2. doi: 10.1016/j.apmr.2006.05.016. PMID 16935068
- [Background] Dibble LE, Hale TF, Marcus RL, Droge J, Gerber JP, LaStayo PC. High-intensity resistance training amplifies muscle hypertrophy and functional gains in persons with Parkinson's disease. Mov Disord. 2006 Sep;21(9):1444-52. doi: 10.1002/mds.20997. PMID 16773643
- [Background] Dibble LE, Hale TF, Marcus RL, Gerber JP, LaStayo PC. High intensity eccentric resistance training decreases bradykinesia and improves Quality Of Life in persons with Parkinson's disease: a preliminary study. Parkinsonism Relat Disord. 2009 Dec;15(10):752-7. doi: 10.1016/j.parkreldis.2009.04.009. Epub 2009 Jun 3. PMID 19497777
- [Result] Foreman KB, Addison O, Kim HS, Dibble LE. Testing balance and fall risk in persons with Parkinson disease, an argument for ecologically valid testing. Parkinsonism Relat Disord. 2011 Mar;17(3):166-71. doi: 10.1016/j.parkreldis.2010.12.007. Epub 2011 Jan 6. PMID 21215674
- [Derived] Dibble LE, Foreman KB, Addison O, Marcus RL, LaStayo PC. Exercise and medication effects on persons with Parkinson disease across the domains of disability: a randomized clinical trial. J Neurol Phys Ther. 2015 Apr;39(2):85-92. doi: 10.1097/NPT.0000000000000086. PMID 25742370